CLINICAL TRIAL: NCT04671745
Title: Qualitative Study of the Effect of Interactive Music on the " Child Centered Care Theory " During Dressing Changes in Children.
Brief Title: MUSIQ: MusicStudyImpactQualitative
Acronym: MUSIQ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201159
Record Dates: First submitted 2020-11-19; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Pain
Keywords: Music; pain; Dressing; Childcentred care; Interaction
MeSH Terms: conditions — Pain | interventions — Music Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Expérimental: patient receiving care with interactive music
  Interventions: Behavioral: Music
- Control: patient receiving care without interactive music
  Interventions: Behavioral: No music

INTERVENTIONS:
Behavioral: Music — patient receiving care with interactive music
  Groups: Expérimental
Behavioral: No music — patient receiving care without interactive music
  Groups: Control

SUMMARY:
Dressing repairs cause distress and pain in children. Although drug analgesia is commonly used, some young children experience pain, distress and agitation.

In these cases, the practice of care is not in line with a child-centred approach (CCC). In addition, the use of non-pharmacological methods is recommended to optimize a child procedural pain management . In addition, the use of non-pharmacological methods is recommended to optimize a child procedural pain management in pediatrics. For this reason, interactive music can be proposed during the course of care. We suggest that interactive music transforms behaviour, attitudes, beliefs and convictions of the child, parents and caregivers during the dressing process, thereby altering the perception of pain and the overall experience of care.

The aim of this qualitative study is to explore what happens when children receive dressings in the presence of a musician trained in interactive music distribution in a hospital. Qualitative data will be generated through observation of clinical procedures by non-participant observers (n25) and semi-structured interviews with the musician, healthcare professionals, parents and children to explore this phenomenon from the participants' perspective. The data will be analysed by constant comparison. We will examine the actions, inactions and interactions of healthcare professionals, parents and children during dressing changes through the central theoretical concept of 'Child Centered Care'.

DETAILED DESCRIPTION:
Pain and distress in children as a result of care procedures is documented (1) (2). Acute pain may have consequences in the short and long term(6) (7) (8,9). According to a Canadian study(10) the prevalence of procedural pain is 78% in the first 24 hours of hospitalization, dressing changes are common and are part of procedures that generate pain, including severe pain.

The influence of distress and anxiety is demontred in the modulation of pain perception (18,19). Therefore, the prevention of procedural pain must be multimodal (20). The value of non-pharmacological means to reduce pain and reduce the distress of the child during procedures is documented. (21-26). These approaches also help to limit the use of restraint during procedure. This practice is strating to be explored in the professional literature (27-32). The hypothesis of "transient empathic blindness" in the use of strong restraint during care " (37) could help to understand what happens in these circumstances. This phenomenon is to be linked to either a child-centred approach or one that focuses on the performance of the procedure. The Child Centered Care Theory suggests that child-centered care should be produced by focusing on the child himself or herself (38,39). These approaches are based on a combination of attitudes and behaviours that adjust to the child's reactions, welcome his emotions, respect his pacing, and allow him to make choices. This observation opens up new perspectives in the way in which the role of non-pharmacological methods is considered, particularly those involving more specifically human interactions. For they allow a practical and effective mediation of the relationship with the child.

According to a review of the literature concerning the effectiveness of integrative approaches to pain and anxiety in children and adolescents with cancer (46), music is one of the main strategies used by paediatric professionals to reduce pain and anxiety in children with distraction, virtual reality, hypno-analgesia, and massage, although the lack of randomized clinical trials concerning the use of these methods is to be deplored.

Randomized clinical trials on the value of music for procedural (23,53,54) or postoperative (55-57) pain have been conducted. There are several modalities for using music in the health field. These may be listening to recorded music (55,58,59) or to a specific programme to be listened to, or listening to so-called interactive music, i.e. a live musical session with the child by a musician (60,61). Interactive (or active) music, i.e., provided by a qualified musician trained in hospital intervention, using voice, body language and facial expression, can involve the child in a way that recorded music cannot (62). A meta-analysis of 30 early studies of the use of music in medical and dental procedures supports this assertion (63). One study compared the effects of live singing and guitar playing on adult patients hospitalized for cancer with the effects of recorded music of the same type. Active music allows for personalized musical expression that can be improvised in the context of care. This can be particularly crucial for young children to feel more comfortable. Indeed, musical support provided by song and an instrument may be best adapted to the child's immediate experience, as well as that of the parents and healthcare professionals providing the treatment. Indeed, we can imagine that music can help to introduce good interaction, which helps to regulate professional relations and relations with the patient and other professionals.

Live music was found to be more effective than recorded music in reducing anxiety and discomfort. (65) It is also known that parental stress can be significant when their child is ill and during medical procedures(68,69). Listening to music can reduce parental stress and improve parent-child interactions(48,70).

(48,70) Based on this finding, interactive music can transform the behaviours, attitudes, beliefs and convictions of the child, parents and caregivers.

Based on this observation, we could imagine that interactive music transforms the behaviours, attitudes, beliefs and convictions of the child, parents and caregivers when performing dressings, thus changing the child's approach and thus his behaviour and perception of treatment and pain. It is proposed that a child-centred approach improves care. The research hypothesis is therefore about the possibility that interactive music may promote a child-centred approach.

To date, no qualitative study has investigated the use of interactive music from the perspective of the participants in the theoretical perspective of the child-centred approach.

Qualitative research could explore what happens when children receive dressings on an outpatient basis in the presence of a musician trained in interactive music distribution at a teaching hospital by generating qualitative data through non-participatory observations of clinical procedures and semi-structured interviews with participants (musicians, health professionals, parents and children).

The aim is to question the triangulation of interactions from a philosophical and political perspective. The originality of this research is to seek to highlight the impact of interactive music on the philosophy of care through the central theoretical concept of "Child Centered Care". More globally, the vocation of this qualitative study is to widen the questioning to the political dimension by questioning the intervention of interactive music (human intervention) as a mediator of the social link. This exploratory qualitative study guided by the principles of grounded theory (71,72) will examine the actions, inactions and interactions that occur throughout the course of dressing changes, with an emphasis on the child's place in the interactions.

ELIGIBILITY:
Inclusion Criteria:

- All children (from 0 to 16 years old) accompanied by their parent who need to have their bandage repaired

Exclusion Criteria:

* Patient known to have severe hearing impairment warranting the use of hearing aids
* Patient with a life-threatening emergency
* End-of-life patient
* Patient not benefiting from social security
* Patient benefiting from State Medical Aid
* Child whose parents are opposed to participation in research
* Parent who does not understand the French language
* Protected adult parents
* Parent or child who refuses the musician's presence

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children (1 to 16 years old) who must have a bandage made with interactive music and who do not meet the criteria for non-inclusion.
  The parents of the children concerned by the observations, present during the care, having a good command of the French language.
  Professionals involved in care Musicians participating in the interactive music program
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
observation grid developed on the basis of the main theoretical axes of CCC (Child Centred Care) | the day of inclusion, up to one week after inclusion
  Observe and record the interactions and behaviours of the child and caregivers during the procedure.

SECONDARY OUTCOMES:
describe and conceptualize the processes involved when health professionals care for and interact with the child in the presence of active music and explain these processes. | the day of inclusion
  collect the words of parents and children to understand their point of view regarding the procedure performed with music
The FLACC (Face Legs Activity Cry Consolability) scale's score. | the day of inclusion
  The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
The PRIC (Procedural Restraint Intensity in Children) scale's score. | the day of inclusion
  The scale is scored in a range of 4 levels
The EVAN (Evaluation of Anxiety) scales's score | the day of inclusion
  The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte LOMBART, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Saint Antoine Coordination générale des soins, Paris, France

IPD SHARING:
Plan to Share IPD: No